CLINICAL TRIAL: NCT02780492
Title: Developing Tools for Assessing the Natural History of Ambulant and Non-ambulant DMD Individuals to Assist in Antisense-oligomer Clinical Trials
Brief Title: Outcome Measures in Duchenne Muscular Dystrophy: A Natural History Study
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other); University of Newcastle Upon-Tyne (Other); Groupe Hospitalier Pitie-Salpetriere (Other); Leiden University Medical Center (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 12/0096 (09DN17)
Record Dates: First submitted 2016-05-19; First posted 2016-05-23 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; Natural history; Outcome measures; North Star Ambulatory Assessment (NSAA); 6 minute walk distance (6MWD); Myoset; Exon skipping
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Single sample suitable for testing for SNP genotyping. This can be either a blood sample, saliva sample or already extracted DNA sample (including stored DNA samples from a laboratory.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Ambulant patients: A set of assessment tools (blood analyses, functional, respiratory, quality of life questionnaires, Dexa scan, MRI) will be performed.
  Interventions: Other: Set of assessment tools
- Non-ambulant patients: A set of assessment tools (blood analyses, functional, respiratory, quality of life questionnaires, Dexa scan, MRI) will be performed.
  Interventions: Other: Set of assessment tools
- Healthy volunteers and Disease controls: A set of assessment tools (upper limb function tests, MRI, blood analyses) will be performed
  Interventions: Other: Set of assessment tools

INTERVENTIONS:
Other: Set of assessment tools

SUMMARY:
Novel emerging therapies for Duchenne Muscular Dystrophy (DMD) require a deeper understanding of DMD natural history. This study aim to assess the natural history of DMD through a composite assessment tool capable of capturing disease progression linking ambulant and non-ambulant phases of the disease.

DETAILED DESCRIPTION:
Novel emerging therapies for Duchenne Muscular Dystrophy (DMD) require a deeper understanding of DMD natural history. This study aim to assess the natural history of DMD through a composite assessment tool capable of capturing disease progression linking ambulant and non-ambulant phases of the disease.

With a recruitment target of 80 DMD patients across 5 centres (London, Newcastle, Paris, Leiden, Nijmegen), subjects are assessed 6 monthly according to a shared protocol. Assessments include 6-minute walk distance (6MWD), North Star Ambulatory Assessment (NSAA), Performance of Upper Limb (PUL) and MyoSet (myogrip, myopinch and moviplate). Both ambulant and non-ambulant subjects undergo upper limb evaluation and respiratory function test including forced vital capacity (FVC), maximum inspiratory and expiratory pressures (MIP/MEP). A subgroup of patients performs annual whole body DEXA scan. An imaging sub-study will aim to characterize muscle (upper/lower limb) and brain MRI.

The investigators will analyze the longitudinal data for the different assessment tools and explore correlations among them.

This study will offer a comprehensive natural history of DMD including novel outcome measures, allowing to capture disease progression and explore the relationship between different assessment tools.

ELIGIBILITY:
Inclusion Criteria:

For non-ambulant patients:

1. Children and teenagers aged between 5 and 18 years with DMD, who have lost the ability to walk 10 meters with no support
2. The diagnosis of DMD must be documented by genetic testing. If a muscle biopsy is available, it should contain less than 10% of revertant fibres
3. Patients should have deletions amenable of skipping of exons 51 or 53 or 45 or 44 or 46 or 50 or 52
4. Patients should be capable of sitting upright in a wheelchair for at least an hour
5. Patients should be stable from a respiratory point of view. Artificial ventilation with either Bipap or tracheostomy is not a contraindication to the study.
6. Informed consent signed by a parent/legal guardian (or by the patient if 16 years of age).
7. In France, a subject will be eligible for inclusion in this study only if either affiliated to, or a beneficiary of, a social security category.

For ambulant patients:

1. Ambulant children from 5 years old and teenagers with DMD, and potential candidates for future genetic therapies with antisense oligomer (AO) exon skipping
2. The diagnosis of DMD must be documented by MLPA or a standard genetic test for the disorder, genotypically confirmed to have an out-of-frame deletion(s) that could be corrected by skipping exon 51 or 53 or 45 or 44 or 46 or 50 or 52
3. If a muscle biopsy is available less than 10% revertant fibres
4. Ability to walk independently for at least 75 meters in 6 minutes at recruitment.
5. Patients should receive the standard of care for DMD as recommended by the NorthStar UK and TREAT-NMD (i.e.: on glucocorticoids treatment)
6. Sufficiently preserved pulmonary function (FVC >30%) and absence of symptoms of cardiac failure
7. Informed consent signed by a parent/legal guardian (or by the patient if 16 years of age)
8. In France, a subject will be eligible for inclusion in this study only if either affiliated to, or a beneficiary of, a social security category.

For healthy volunteers and disease controls:

1. Participant are able to provide informed consent/assent for taking blood samples and/or performing limb MRI and/or physiotherapy assessment of the upper limb function
2. Participants have a neuromuscular disease that is not Duchenne Muscular Dystrophy or are a healthy volunteer with no neuromuscular disease
3. Able to have a blood sample taken

Exclusion Criteria:

For non-ambulant patients:

1. Patients who are currently involved in interventional clinical trials aimed at restoring dystrophin will be excluded, as their data could not be used to establish natural history of the disease (participation in a previous interventional clinical trial prior to 6 months from being recruited in the study is not an exclusion criterion)
2. Patients with severe intellectual impairment, who would be unable to cooperate with examination
3. Patients/families the investigators anticipate may have emotional/ psychological problems if recruited into a natural history study
4. Symptomatic cardiac failure
5. Recent (< 6 months) upper limb surgery or trauma
6. Anticipated surgery for anytime during the duration of the study
7. None of the current treatments for DMD are exclusion criteria
8. For the MRI sub-study, patients with metal/metallic surgically inserted equipment incompatible with MRI scan will be excluded as well as patients suffering from claustrophobia.

For ambulant patients:

1. Patients who are currently involved in interventional clinical trials aimed at restoring dystrophin will be excluded, as their data could not be used to establish natural history of the disease (participation in a previous interventional clinical trial prior to 6 months from being recruited in the study is not an exclusion criterion)
2. Patients with severe intellectual impairment, who would be unable to cooperate with examination
3. Patients/families the investigators anticipate may have emotional/ psychological problems if recruited into a natural history study
4. Recent surgery or anticipated for anytime during the duration of the study
5. For the MRI sub-study, patients with metal/metallic surgically inserted equipment incompatible with MRI scan will be excluded as well as patients suffering from claustrophobia.

For healthy volunteers and disease controls

1. Patients who are currently involved in interventional clinical trials aimed at restoring dystrophin will be excluded, as their data could not be used to establish natural history of the disease (participation in a previous interventional clinical trial prior to 6 months from being recruited in the study is not an exclusion criterion)
2. Patients with severe intellectual impairment, who would be unable to cooperate with examination
3. Patients/families the investigators anticipate may have emotional/ psychological problems if recruited into a natural history study
4. For the MRI sub-study, patients with metal/metallic surgically inserted equipment incompatible with MRI scan will be excluded as well as patients suffering from claustrophobia

Ages: 5 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with Duchenne muscular dystrophy (DMD) recruited across 5 specialised neuromuscular centres (London, Newcastle, Paris, Leiden, Nijmegen)
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2012-04-11 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Disease progression | up to 4 years
  Evaluate disease progression from ambulant to non-ambulant patients through a composite assessment tool

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Muntoni, PhD, Principal Investigator — Dubowitz Neuromuscular Centre, UCL-Institute of Child Health
Locations (5):
- Institut de Myologie, Groupe Hospitalier Pitié Salpêtrière, Paris, France
- Netherlands (2):
  - Leiden University Medical Centre, Leiden
  - Radboud University Medical Centre, Nijmegen
- United Kingdom (2):
  - Dubowitz Neuromuscular Centre, UCL-Institute of Child Health, London
  - John Walton Muscular Dystrophy Research Centre, Newcastle University, Newcastle

IPD SHARING:
Plan to Share IPD: Yes
The results of the study will be published in peer-reviewed scientific journal(s), presented at relevant national and international meetings and reported as part of submissions to regulatory bodies (NHS R&D offices and Research Ethics Committee).
Supporting Information: Study Protocol
Time Frame: Up to five years
Access Criteria: Researchers to obtain permission from the study team.

REFERENCES:
- [Derived] Ayyar Gupta V, Pitchforth JM, Domingos J, Ridout D, Iodice M, Rye C, Chesshyre M, Wolfe A, Selby V, Mayhew A, Mazzone ES, Ricotti V, Hogrel JY, Niks EH, de Groot I, Servais L, Straub V, Mercuri E, Manzur AY, Muntoni F; iMDEX Consortium and the U.K. NorthStar Clinical Network. Determining minimal clinically important differences in the North Star Ambulatory Assessment (NSAA) for patients with Duchenne muscular dystrophy. PLoS One. 2023 Apr 26;18(4):e0283669. doi: 10.1371/journal.pone.0283669. eCollection 2023. PMID 37099511
- [Derived] Trucco F, Ridout D, Domingos J, Maresh K, Chesshyre M, Munot P, Sarkozy A, Robb S, Quinlivan R, Riley M, Wallis C, Chan E, Abel F, De Lucia S, Hogrel JY, Niks EH, de Groot I, Servais L, Straub V, Ricotti V, Manzur A, Muntoni F; UK NorthStar Clinical Network and AFM Network. Genotype-related respiratory progression in Duchenne muscular dystrophy-A multicenter international study. Muscle Nerve. 2022 Jan;65(1):67-74. doi: 10.1002/mus.27427. Epub 2021 Oct 27. PMID 34606104
- [Derived] Catapano F, Scaglioni D, Maresh K, Ala P, Domingos J, Selby V, Ricotti V, Phillips L, Servais L, Seferian A, Groot I, Krom YD, Voit T, Verschuuren JJGM, Niks EH, Straub V, Morgan J, Muntoni F. Novel free-circulating and extracellular vesicle-derived miRNAs dysregulated in Duchenne muscular dystrophy. Epigenomics. 2020 Nov;12(21):1899-1915. doi: 10.2217/epi-2020-0052. Epub 2020 Nov 20. PMID 33215544